CLINICAL TRIAL: NCT06652308
Title: Frequency of Unipolar and Bipolar Mood Disorders in Patients with Multiple Sclerosis: a Retrospective Cohort Study
Brief Title: Mood Disorders in Multiple Sclerosis Patients
Acronym: MSMD
Status: Completed | Type: Observational
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Shaghayegh Radmehr, Dr, Islamic Azad University, Sanandaj
Other Study IDs: MSMood2024-SDU
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis (MS); Unipolar Depression; Bipolar Disorder; Mood Disorders
Keywords: Multiple Sclerosis; Mood Disorders; Unipolar Depression; Mental Health
MeSH Terms: conditions — Multiple Sclerosis; Depressive Disorder; Bipolar Disorder; Mood Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple Sclerosis Patients with Mood Disorders

SUMMARY:
This study investigates the frequency of unipolar and bipolar mood disorders in patients with multiple sclerosis. MS is a chronic condition that affects the central nervous system, and previous research suggests that mood disorders, such as depression and bipolar disorder, may occur more frequently in MS patients compared to the general population.

A retrospective analysis of 85 patients diagnosed with MS was conducted, evaluating lifetime experiences with mood disorders using structured clinical interviews. The goal is to better understand the prevalence of these mood disorders and to raise awareness of the importance of mental health care in patients with MS. The findings highlight that mood disorders, particularly bipolar disorder, are more common in MS patients than previously thought. This information can help healthcare providers improve screening, diagnosis, and treatment for MS patients suffering from mood disorders.

DETAILED DESCRIPTION:
This study is a retrospective cohort analysis designed to examine the lifetime prevalence of unipolar and bipolar mood disorders in patients with multiple sclerosis. MS is a chronic, demyelinating condition of the central nervous system that leads to varying degrees of neurological impairment. Previous studies have shown that mood disorders, particularly depression and bipolar disorder, are more prevalent in patients with MS than in the general population.

Data from 85 patients (45 females and 40 males) diagnosed with MS were analyzed, focusing on psychiatric history through structured clinical interviews. The study evaluated the presence of mood disorders, including major depressive disorder, bipolar disorder types I and II, dysthymia, and unclassified mood disorders. Data were collected using DSM-IV criteria to ensure consistency in diagnosis.

The results demonstrate that mood disorders, especially bipolar disorder, are more frequent than previously reported in this patient population. These findings underscore the need for improved mental health screening and treatment for MS patients, as managing psychiatric comorbidities can significantly enhance overall quality of life. The study emphasizes the importance of integrating psychiatric care into routine MS management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis: Participants must have a confirmed diagnosis of multiple sclerosis (MS) by a qualified neurologist.
* Age Range: Participants must be between 18 and 65 years of age.
* Informed Consent: Participants must provide informed consent to participate in the study.
* Geographic Location: Participants must reside in Tehran, Iran.

Exclusion Criteria:

* Other Neurological Disorders: Individuals with a diagnosis of any other neurological disease (e.g., epilepsy, Parkinson's disease) will be excluded.
* Head Trauma: History of head trauma that resulted in impaired consciousness or memory loss.
* Seizures: A history of seizures that could affect mood.
* Substance Dependence: A history of substance dependence as per DSM-IV criteria.
* Other Physical Illnesses: Any systemic or physical diseases that could lead to mood symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 85 patients diagnosed with multiple sclerosis who were selected through simple random sampling from the Iranian MS Association. The cohort includes:
  Gender Distribution:
  45 females (52.9%) 40 males (47.1%)
  Age Range:
  Participants are aged between 18 and 65 years. The average age of participants is approximately 5.47 years (please verify if this is correct as it seems like it might be a typo).
  Geographic Location:
  All participants reside in Tehran, Iran.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
6-year Frequency of Mood Disorders | 6-year assessment (from diagnosis of MS).
  The primary outcome measure is the 6-year frequency of mood disorders (unipolar and bipolar) diagnosed in patients with multiple sclerosis (MS). This will be evaluated using semi-structured clinical interviews based on DSM-IV criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: No